CLINICAL TRIAL: NCT05476211
Title: Safety and Efficacy of the BTL-785F Device for Non-invasive Reduction of Wrinkles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-785_CTBG100
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Wrinkle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Reduction of wrinkles (Experimental)
  Interventions: Device: BTL-785F

INTERVENTIONS:
Device: BTL-785F — Radiofrequency

SUMMARY:
This study will evaluate the clinical safety and the performance of the BTL-785F system for non-invasive treatment of facial wrinkles. The study is a multicenter single-arm, open-label, interventional study. The subjects will be enrolled and assigned into one experimental study arm. The subjects will be required to complete four (4) treatment visits and two follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects over 21 years of age seeking treatment for reduction of wrinkles
* Subjects should be able understand the investigative nature of the treatment, the possible benefits and side effects, and must sign the Informed Consent Form
* Presence of clearly visible wrinkles in the treated areas (forehead, cheeks) when the face is relaxed as deemed appropriate by the Investigator
* Subjects willing and able to abstain from partaking in any facial treatments other than the study procedure during study participation
* Willingness to comply with study instructions, to return to the clinic for the required visits, and to have photographs of their face taken

Exclusion Criteria:

* Local bacterial or viral infection in the area to be treated
* Local acute inflammation in the area to be treated
* Impaired immune system caused by any immunosuppressive illness, disease or medication
* Isotretinoin and tretinoin-containing medication use in the past 12 months
* Skin related autoimmune diseases
* Radiation therapy and/or chemotherapy
* Poor healing and unhealed wounds in the treatment area
* Metal implants
* Permanent implant in the treated area
* Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body
* Facial dermabrasion, facial resurfacing, or deep chemical peeling in the treatment area within 3 months prior to the treatment
* Current or history of skin cancer, or current condition of any other type of cancer, or pre-malignant moles
* History of skin disorders, keloids, abnormal wound healing and dry or fragile skin
* History of any type of cancer
* Active collagen diseases
* Cardiovascular diseases (such as vascular diseases, peripheral arterial disease, thrombophlebitis and thrombosis)1
* Pregnancy/nursing or IVF procedure
* History of bleeding coagulopathies, use of anticoagulants
* Any active condition in the treatment area, such as sores, psoriasis, eczema, rash and rosacea
* Any surgical procedure in the treatment area within the last three months or before complete healing
* Poorly controlled endocrine disorders, such as diabetes
* Acute neuralgia and neuropathy
* Kidney or liver failure
* Nerve insensitivity (sensitivity disorders) to heat in the treatment area
* Varicose veins, pronounced edemas1
* Prior use of dermal fillers, botulinum toxin, lasers, etc. therapies in the treated area that can influence the study results at the investigator discretion
* Unwillingness/inability to not change their usual cosmetics and especially not to use anti-aging or anti-wrinkles products in the treated area during the duration of the study including the follow-up period
* Electroanalgesia without exact diagnosis of pain etiology
* Neurological disorders (such as multiple cerebrospinal sclerosis, epilepsy)
* Blood vessels and lymphatic vessels inflammation
* Any other disease or condition at the investigator discretion that may pose risk to the patient or compromise the study

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Assess reduction of wrinkle severity according to the Fitzpatrick Wrinkle and Elastosis Scale | 4 months
  The primary efficacy outcome measure is a statistically significant reduction of at least 1.0 score in the average score of Fitzpatrick Wrinkle and Elastosis Scale score according to at least 2 out of 3 blinded dermatologists at 3-months follow-up compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for specialized medical care - Individual dermatological practice Dr. Mariya Genova, Plovdiv, Bulgaria

IPD SHARING:
Plan to Share IPD: No